CLINICAL TRIAL: NCT00816127
Title: Intranasal DDAVP in Preventing Bleeding During Dental Extraction in Cirrhotic Patients
Brief Title: Prevention of Bleeding in Patient With Cirrhosis Undergoing Dental Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Thomas D. Schiano, M.D, Mount Sinai School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-0727
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Liver Cirrhosis; Coagulopathy
Keywords: liver cirrhosis; coagulopathy; desmopressin; blood transfusion
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders | interventions — Deamino Arginine Vasopressin; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DDAVP
  Interventions: Drug: Desmopressin
- 2 (Active Comparator): Standard Treatment
  Interventions: Biological: blood transfusion

INTERVENTIONS:
Drug: Desmopressin — intranasal desmopressin (300μg)
  Arms: 1
Biological: blood transfusion — fresh frozen plasma 10ml/kg and/or 1 unit of single donor platelets
  Arms: 2

SUMMARY:
The purpose of this study is to investigate how effective and cost saving 1-deamino-8-D-arginine vasopressin (desmopressin, DDAVP) is as opposed to the transfusion of blood products in preventing bleeding after teeth extraction in persons with severe liver disease being evaluated for liver transplant.

DETAILED DESCRIPTION:
Liver cirrhosis is associated with dysregulation of the coagulation system resulting in an increased bleeding tendency in cirrhotic patients. The treatment approach to offset these abnormalities may involve transfusion with fresh frozen plasma (FFP) and platelets. Fluid overload may become a concern as the large amount of FFP (10-20mls/kg or >1,500ml) required to achieve the hemostatic effect could be contraindicated in some patients. Furthermore, repeated platelet transfusion induces alloimmunization and refractoriness to new transfusion, which is an important issue in patients on the waiting list for liver transplantation in which HLA-matched and cross-matched platelets may be required. Non-transfusional drugs that help to stop bleeding have been used in patients with congenital bleeding disorders. 1-deamino-8-D-arginine vasopressin (DDAVP, Desmopressin), a synthetic analogue of the antidiuretic hormone, L-arginine, has been used as a non-transfusional form of replacement therapy in a variety of congenital and acquired bleeding disorders. Through unknown mechanisms, DDAVP shortens the prolonged bleeding times of cirrhotic patients despite the high plasma concentrations of Factor VIII and von Willebrand factor sound in chronic liver disease, indicating that it might be useful as a prophylactic treatment in cirrhotic patients undergoing minimally invasive procedures, i.e. dental extraction.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with biopsy-proven liver cirrhosis or clinical/radiological evidence of cirrhosis, requiring dental extraction
* platelet count of 30,000-50,000/microL and/or INR 2.0-3.0

Exclusion Criteria:

* the presence of other bleeding disorders besides cirrhosis such as renal dysfunction (creatinine > 2.0) or HIV
* receipt of blood transfusion within 2 weeks prior to study
* recent acute decompensation of liver cirrhosis
* malignancy excluding hepatocellular carcinoma in the absence of portal vein thrombosis
* treatment with anti-platelet medications (aspirin, non-steroidal anti-inflammatory drugs or clopidogrel) within ten days prior to the extraction
* documented allergy to DDAVP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Necessity of rescue blood transfusion in patients who received DDAVP or blood transfusion prior to dental extraction. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D. Schiano, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Amitrano L, Guardascione MA, Brancaccio V, Balzano A. Coagulation disorders in liver disease. Semin Liver Dis. 2002 Feb;22(1):83-96. doi: 10.1055/s-2002-23205. PMID 11928081
- [Background] Kobrinsky NL, Israels ED, Gerrard JM, Cheang MS, Watson CM, Bishop AJ, Schroeder ML. Shortening of bleeding time by 1-deamino-8-D-arginine vasopressin in various bleeding disorders. Lancet. 1984 May 26;1(8387):1145-8. doi: 10.1016/s0140-6736(84)91393-x. PMID 6144876
- [Background] de la Fuente B, Kasper CK, Rickles FR, Hoyer LW. Response of patients with mild and moderate hemophilia A and von Willebrand's disease to treatment with desmopressin. Ann Intern Med. 1985 Jul;103(1):6-14. doi: 10.7326/0003-4819-103-1-6. PMID 3923887
- [Background] Mannucci PM, Remuzzi G, Pusineri F, Lombardi R, Valsecchi C, Mecca G, Zimmerman TS. Deamino-8-D-arginine vasopressin shortens the bleeding time in uremia. N Engl J Med. 1983 Jan 6;308(1):8-12. doi: 10.1056/NEJM198301063080102. PMID 6401193
- [Background] Saulnier J, Marey A, Horellou MH, Goudemand J, Lepoutre F, Donazzan M, Gazengel C, Torchet M, Letang C, Schuhmann C, et al. Evaluation of desmopressin for dental extractions in patients with hemostatic disorders. Oral Surg Oral Med Oral Pathol. 1994 Jan;77(1):6-12. doi: 10.1016/s0030-4220(06)80099-x. PMID 8108099
- [Background] Mannucci PM, Ruggeri ZM, Pareti FI, Capitanio A. 1-Deamino-8-d-arginine vasopressin: a new pharmacological approach to the management of haemophilia and von Willebrands' diseases. Lancet. 1977 Apr 23;1(8017):869-72. doi: 10.1016/s0140-6736(77)91197-7. PMID 67283
- [Background] Mannucci PM. Desmopressin (DDAVP) in the treatment of bleeding disorders: the first 20 years. Blood. 1997 Oct 1;90(7):2515-21. No abstract available. PMID 9326215